CLINICAL TRIAL: NCT05834023
Title: Comparison Between Bupivacaine 0.5% Versus Bupivacaine 0.25% Plus Lidocaine 1% in Ultrasound-guided Infraclavicular Block: a Prospective Randomized Controlled Trial
Brief Title: Bupivacaine Versus Bupivacaine Plus Lidocaine in Infraclavicular Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de San Carlos Dr. Benicio Arzola Medina (Other)
Responsible Party: Principal Investigator, Germán Armando Aguilera Ceballos, Principal Investigator, Hospital de San Carlos Dr. Benicio Arzola Medina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CEC-HCHM 05-2023
Record Dates: First submitted 2023-04-06; First posted 2023-04-27 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Pain, Acute; Postoperative Pain; Analgesia
Keywords: Bupivacaine; Lidocaine; Nerve Block; Infraclavicular Block; Upper Extremity Surgery
MeSH Terms: conditions — Acute Pain; Pain, Postoperative; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A research assistant will prepare the solutions before the procedure, utilizing bupivacaine alone or mixing bupivacaine and lidocaine as appropriate. The operator, patient, and investigator assessing the block will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine 0.25% plus Lidocaine 1% (Active Comparator): Infraclavicular block with Bupivacaine and Lidocaine
  Interventions: Drug: Bupivacaine-Lidocaine
- Bupivacaine 0.5% (Experimental): Infraclavicular block with Bupivacaine
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine-Lidocaine — Infraclavicular block with 35 ml of the following anesthetic solution: Bupivacaine 0.25% + Lidocaine 1% + dexamethasone 4 mg + epinephrine 5 mcg/ml
  Arms: Bupivacaine 0.25% plus Lidocaine 1%
Drug: Bupivacaine — Infraclavicular block with 35 ml of the following anesthetic solution: Bupivacaine 0.5% + dexamethasone 4 mg + epinephrine 5 mcg/ml
  Arms: Bupivacaine 0.5%

SUMMARY:
In this study, the investigators will compare two different anesthetic solutions in the infraclavicular block in patients having forearm, wrist, and hand surgery. The solutions will be bupivacaine 0.5% versus bupivacaine 0.25% plus lidocaine 1%, both associated with epinephrine 5 mcg/ml and dexamethasone 4 mg.

The main objective of this investigation is to demonstrate that using higher concentrations of bupivacaine alone results in a significant block duration increase compared with the mixture of bupivacaine and lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* American Society of Anesthesiologists classification 1-3
* Surgery of the forearm, wrist, and hand
* Weight ≥ 80 kilograms

Exclusion Criteria:

* Adults who are unable to give their consent
* Infection in the injection site (infraclavicular region)
* Pre-existing neuropathy (assessed by history and physical examination)
* Coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work, i.e., platelets ≤ 100, International Normalized Ratio ≥ 1.4)
* Renal failure (assessed by history and physical examination and if deemed clinically necessary, by blood work, i.e., creatinine ≥ 1.2)
* Hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work, i.e., transaminases ≥ 100)
* Allergy to local anesthetics (LAs)
* Pregnancy or breastfeeding
* Prior surgery in the infraclavicular region
* Chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Motor block duration | 0 - 48 hours after block
  The time interval in minutes between the end of the local anesthetic injection and the return of hand mobility.

SECONDARY OUTCOMES:
Sensory block duration | 0 - 48 hours after block
  The time interval in minutes between the end of the local anesthetic injection and the return of hand sensation.
Analgesic block duration | 0 - 48 hours after block
  The time interval in minutes between the end of the local anesthetic injection and the first sensation of pain in the surgical area.
Sensory and motor block score | 0 - 60 minutes after block
  The sensorimotor block will be assessed every 5 minutes until 60 minutes after the end of local anesthetic injection using a 16-point composite score evaluating sensory and motor block of musculocutaneous, median, radial, and ulnar nerves.
  Sensation will be assessed with a pinprick test in each nerve territory with a 0 to 2-point scale. 0= no block, patients can feel a pin prick; 1= analgesic block, the patient can feel touch but not pinprick; 2= anesthetic block, the patient cannot feel pinprick or touch.
  The motor function will be assessed for each nerve with a 0 to 2 points scale where 0= no motor block; 1= paresis; 2= paralysis.
Block onset time | 0 - 60 minutes after block
  The time interval in minutes between the end of the local anesthetic injection and a minimal sensorimotor composite score of 14 out of 16 points.
  The sensorimotor score is described in Outcome 4.
Incidence of successful block | 0 - 60 minutes after block
  Patients with a minimal sensorimotor score of 14 out of 16 points, with at least 7 points in the sensitive score. The sensorimotor score is described in Outcome 4.
Incidence of failed block | 0 - 60 minutes after block
  Patients with a sensorimotor score of 13 points or less. The sensorimotor score is described in Outcome 4.
Incidence of anesthetic block | 60 to 120 minutes after the ending time of local anesthetic injection
  Ability to proceed with the surgery without general anesthesia, rescue blocks, or local anesthesia infiltration by the surgeon.
Procedural pain | Immediately after nerve block
  Pain related to the nerve block according to the Numeric Rating Scale for Pain. This scale is graduated from 0 to 10 points. A 0-point score represents the absence of pain, and a 10-point score means the worst imaginable pain.
Image time | 2 hours before surgery
  The time interval in seconds between the probe placement and the acquisition of the final ultrasonographic image.
Needle time | 2 hours before surgery
  The time interval in seconds between the skin infiltration and the end of local anesthetic injection
Block performance time | 2 hours before surgery
  Sum of image and needle time
Number of patients requiring general anesthesia | 60 to 120 minutes after the ending time of local anesthetic injection
  Patients who need general anesthesia to proceed with the surgery
Diaphragmatic function | From arrival to the pre-anesthesia unit to the end of surgery
  Diaphragmatic excursion in millimeters evaluated by ultrasound in three different times: pre-block, 60 minutes after block, and at the end of the surgery
Rate of diaphragmatic paresis | From 60 minutes after block to the end of the surgery
  Patients with decreased diaphragmatic excursion by 25% to 75% compared with the basal function 60 minutes after the block or at the end of the surgery.
Rate of diaphragmatic paralysis | From 60 minutes after block to the end of the surgery
  Patients with decreased diaphragmatic excursion greater than 75% compared with the basal function, absence of diaphragmatic movement, or paradoxical movement 60 minutes after the block or at the end of the surgery.
Incidence of rebound pain | 24 hours after the block wears off
  Severe pain (NRS ≥ 7) in the surgical area within 24 hours after the block wears off.
Incidence of nerve block side effects | From skin anesthesia to 60 minutes after the nerve block
  The presence of Horner syndrome, paresthesia, vascular puncture, hematoma, or local anesthetic systemic toxicity after the nerve block.
Postoperative complications | 7 days after surgery
  Presence of persistent paresthesia, numbness, or motor deficit in the postoperative period.
Duration of surgery | 3 hours after skin incision
  Time in minutes between skin incision and closure.
Pain score in the post-anesthesia care unit (PACU) | 3 hours after the end of the surgery
  Highest pain reported by the patient in the PACU according to the Numeric Rating Scale for Pain. This scale is graduated from 0 to 10 points. A 0-point score represents the absence of pain, and a 10-point score means the worst imaginable pain.
Length of PACU stay | 3 hours after the end of the surgery
  The time interval in minutes between PACU arrival to readiness to discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de San Carlos Dr. Benicio Arzola Medina, San Carlos, Región de Ñuble, Chile

REFERENCES:
- [Background] Vrancken D, Theunissen M, Joosten EA, Fiddelers AAA, Hoofwijk DMN, Buhre WFFA, Gramke HF, Stessel BOR. Procedure-Specific Pain Intensity Four Days After Day Surgery and the Relationship with Preoperative Pain: A Prospective Cohort Study. Anesth Pain Med. 2018 Nov 17;8(6):e81366. doi: 10.5812/aapm.81366. eCollection 2018 Dec. PMID 30719413
- [Background] Ilfeld BM. Continuous Peripheral Nerve Blocks: An Update of the Published Evidence and Comparison With Novel, Alternative Analgesic Modalities. Anesth Analg. 2017 Jan;124(1):308-335. doi: 10.1213/ANE.0000000000001581. PMID 27749354
- [Background] Aguirre J, Del Moral A, Cobo I, Borgeat A, Blumenthal S. The role of continuous peripheral nerve blocks. Anesthesiol Res Pract. 2012;2012:560879. doi: 10.1155/2012/560879. Epub 2012 Jun 18. PMID 22761615
- [Background] Chelly JE, Ghisi D, Fanelli A. Continuous peripheral nerve blocks in acute pain management. Br J Anaesth. 2010 Dec;105 Suppl 1:i86-96. doi: 10.1093/bja/aeq322. PMID 21148658
- [Background] Sinatra RS, Goldstein R, Sevarino FB. The clinical effectiveness of epidural bupivacaine, bupivacaine with lidocaine, and bupivacaine with fentanyl for labor analgesia. J Clin Anesth. 1991 May-Jun;3(3):219-24; discussion 214-5. doi: 10.1016/0952-8180(91)90164-i. PMID 1878235
- [Background] Ribotsky BM, Berkowitz KD, Montague JR. Local anesthetics. Is there an advantage to mixing solutions? J Am Podiatr Med Assoc. 1996 Oct;86(10):487-91. doi: 10.7547/87507315-86-10-487. PMID 8918026
- [Background] Nestor CC, Ng C, Sepulveda P, Irwin MG. Pharmacological and clinical implications of local anaesthetic mixtures: a narrative review. Anaesthesia. 2022 Mar;77(3):339-350. doi: 10.1111/anae.15641. Epub 2021 Dec 14. PMID 34904711
- [Background] Gadsden J, Hadzic A, Gandhi K, Shariat A, Xu D, Maliakal T, Patel V. The effect of mixing 1.5% mepivacaine and 0.5% bupivacaine on duration of analgesia and latency of block onset in ultrasound-guided interscalene block. Anesth Analg. 2011 Feb;112(2):471-6. doi: 10.1213/ANE.0b013e3182042f7f. Epub 2010 Dec 14. PMID 21156983
- [Background] Bobik P, Kosel J, Swirydo P, Talalaj M, Czaban I, Radziwon W. Comparison of the pharmacological properties of 0.375% bupivacaine with epinephrine, 0.5% ropivacaine and a mixture of bupivacaine with epinephrine and lignocaine - a randomized prospective study. J Plast Surg Hand Surg. 2020 Jun;54(3):156-160. doi: 10.1080/2000656X.2020.1720999. Epub 2020 Jan 31. PMID 32003278
- [Background] Laur JJ, Bayman EO, Foldes PJ, Rosenquist RW. Triple-blind randomized clinical trial of time until sensory change using 1.5% mepivacaine with epinephrine, 0.5% bupivacaine, or an equal mixture of both for infraclavicular block. Reg Anesth Pain Med. 2012 Jan-Feb;37(1):28-33. doi: 10.1097/AAP.0b013e318236bc30. PMID 22157740
- [Background] Almasi R, Rezman B, Kriszta Z, Patczai B, Wiegand N, Bogar L. Onset times and duration of analgesic effect of various concentrations of local anesthetic solutions in standardized volume used for brachial plexus blocks. Heliyon. 2020 Sep 2;6(9):e04718. doi: 10.1016/j.heliyon.2020.e04718. eCollection 2020 Sep. PMID 32944664
- [Background] Pongraweewan O, Inchua N, Kitsiripant C, Kongmuang B, Tiwirach W. Onset Time of 2% Lidocaine and 0.5% Bupivacaine Mixture versus 0.5% Bupivacaine Alone using Ultrasound and Double Nerve Stimulation for Infraclavicular Brachial Plexus Anesthesia in ESRD Patients Undergoing Arteriovenous Fistula Creation. J Med Assoc Thai. 2016 May;99(5):589-95. PMID 27501616
- [Background] Choi S, Rodseth R, McCartney CJ. Effects of dexamethasone as a local anaesthetic adjuvant for brachial plexus block: a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2014 Mar;112(3):427-39. doi: 10.1093/bja/aet417. Epub 2014 Jan 10. PMID 24413428
- [Background] Chong MA, Berbenetz NM, Lin C, Singh S. Perineural Versus Intravenous Dexamethasone as an Adjuvant for Peripheral Nerve Blocks: A Systematic Review and Meta-Analysis. Reg Anesth Pain Med. 2017 May/Jun;42(3):319-326. doi: 10.1097/AAP.0000000000000571. PMID 28252523
- [Background] Desai N, Albrecht E, El-Boghdadly K. Perineural adjuncts for peripheral nerve block. BJA Educ. 2019 Sep;19(9):276-282. doi: 10.1016/j.bjae.2019.05.001. Epub 2019 Jul 6. No abstract available. PMID 33456903
- [Derived] Aguilera G, Tabilo C, Jara A, Aliste J. 0.25% bupivacaine-1% lidocaine vs 0.5% bupivacaine for ultrasound-guided infraclavicular brachial plexus block: a randomized controlled trial. Reg Anesth Pain Med. 2025 Aug 5;50(8):627-634. doi: 10.1136/rapm-2024-105511. PMID 38754989